CLINICAL TRIAL: NCT00493987
Title: The Role of 5-alpha Reductase in Mediating Testosterone Actions
Acronym: 5aR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Dr. Shalender Bhasin, Boston University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HD043348 (NIH); R01HD043348 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Testosterone; Androgens; Dihydrotestosterone; 5-alpha reductase; Body Composition; Muscle; Sexual function; Men; Healthy Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — testosterone enanthate; Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Testosterone enanthate (Active Comparator)
  Interventions: Drug: Testosterone Enanthate
- Duatesteride (Placebo Comparator): Duatesteride
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Testosterone Enanthate — testosterone ester
  Arms: Testosterone enanthate
Drug: Dutasteride — 5 alpha-reductase inhibitor
  Arms: Duatesteride

SUMMARY:
In normal men, the male hormone testosterone affects a number of things in the body including muscle function and sexual function. An enzyme in the body called 5-alpha reductase converts testosterone into another form called dihydrotestosterone (DHT) which has slightly different effects. The purpose of this study is to find out how different amounts of the two different forms of testosterone affect muscle function and sexual function in healthy young men like you. This will be done by giving the men participating in the study different combinations of hormone-related medication for 20 weeks and making measurements before, during and after the medications to look for changes in lean body tissue, muscle size, muscle strength and leg power, as well as sexual function and sexual activity in all participants.

DETAILED DESCRIPTION:
Testosterone, the predominant circulating androgen in men, also serves as a prohormone that is converted in the body to two active metabolites, estradiol 17 β and 5-α DHT (DHT). Testosterone serves as the active hormone in some target tissues; however, androgen effects in other target organs require its conversion to estradiol or DHT. The role of 5-α reduction of testosterone in mediating its effects on the muscle and sexual function remains unclear. Therefore, the primary objective of this project is to determine whether 5-α reduction of testosterone to DHT is obligatory for mediating its effects on fat-free mass, muscle size, muscle strength, and leg power in men. The secondary objective is to determine whether 5-α reduction of testosterone is necessary for maintenance of androgen effects on sexual function (sexual desire, overall sexual activity, nocturnal penile tumescence (NPT), response to visual erotic stimulus, and penile rigidity) in men. In order to test these hypotheses about the role of 5-α reduction, we will compare testosterone dose response curves for each outcome measure in the absence and presence of a novel, potent 5-α reductase inhibitor (dutasteride) that inhibits both type 1 and type 2 steroid 5-α -reductase isoenzymes. Healthy young men, 21-40 years of age, will be treated with a long acting GnRH agonist to suppress endogenous testosterone production, and concomitantly, randomly assigned to one of 8 groups: group 1, testosterone enanthate (TE) 50-mg weekly, plus placebo tablets daily; group 2, TE 125-mg weekly plus placebo daily; group 3, TE 300-mg weekly plus placebo daily; group 4, TE 600 mg TE weekly plus placebo; group 5, 50-mg weekly, plus dutasteride 2.5-mg daily; group 6, TE 125-mg weekly, plus dutasteride daily; group 7, TE 300 mg weekly, plus dutasteride daily; group 8, 600-mg TE plus dutasteride daily. Energy and protein intake, and exercise stimulus will be standardized. The following outcomes will be measured at baseline and after 20 weeks: body composition by DEXA scan, deuterium oxide and sodium bromide dilution; thigh muscle volume by MRI scan; muscle performance by measurements of 1-repetition maximum strength and leg power; sexual function by International Index of Erectile Function, Sexual Desire Inventory, and daily logs of sexual activity; and penile erections and rigidity during EEG-coupled, NPT recoding and in response to a visual erotic stimulus; total and free testosterone, DHT, estradiol, SHBG, and LH levels. For safety, we will follow hemoglobin/hematocrit, sleep apnea scores, AST and ALT, PSA, plasma lipids, apolipoproteins, and lipoprotein particles, and prostate examinations. A multi-disciplinary team of investigators, the use of a previously validated "Leydig Cell Clamp" model, the use of a potent inhibitor of both subtypes of 5-alpha reductase enzyme, attention to potential confounding variables such as energy intake and exercise stimulus, and power and effect size should help elucidate the role of 5-alpha reduction in mediating androgen action. This study will enhance our understanding of the biologic role of the steroid 5-alpha-reductase system, and has immediate clinical relevance in establishing whether selective androgen receptor modulators that do not undergo 5-alpha reduction would be useful as anabolic agents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 18 and 50 years of age.
* Ambulatory, physically active, but not in competitive sports.
* Eugonadal: Normal Serum Testosterone (300-1100 nmol/L).
* Normal LH
* Normal FSH
* Able and willing to comply with the trial protocol.

Exclusion Criteria:

* Known to have a primary or secondary hypogonadism? (e.g. pituitary disease, HIV infection, Klinefelter's Syndrome)
* BMI > 35
* Disability that precludes participation in exercise testing
* Alcohol or illicit drug use in the preceding 6 months that would interfere with participation and compliance with the protocol
* Known disorder that would be exacerbated by androgen treatment e.g. benign prostate hyperplasia, prostate Ca, erythrocytosis, sleep apnea)
* Any abnormalities in the following laboratory tests PSA > 4 ng/ml AST, ALT or Alkaline Phosphatase > 3x ULN? Creatinine level > 2 mg/dL Hematocrit > 51%
* Osteoporosis by DEXA BMD T-Score < -2.5
* Use of medications that affect muscle or bone metabolism within the previous 3 months ?(e.g. glucocorticoids, growth hormone, androgenic steroids, oral androgen precursors -i.e. androstenedione or DHEA)
* Use of medications that affect androgen metabolism, action or clearance within the previous 3 months? (e.g. dilantin, phenobarbital, aldactone, flutamide, finasteride and Ketoconazole)
* Use of ketoconazole or other potent CYP3A4 inhibitors that may affect clearance of dutasteride
* Use investigational medication as part of a research study in the last 3 months?

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2002-11; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fat-free mass, measured by DEXA scanning | 20 weeks

SECONDARY OUTCOMES:
Body composition by Deuterium dilution method | 20 weeks
Maximal voluntary strength in the leg press and chest press exercises. | 20 weeks
Upper and lower extremity muscle power | 20 weeks
Muscle volume by MRI scan | 20 weeks
Prostate volume by MRI Scan | 20 weeks
International Index of Erectile Function | 20 weeks
Men's Sexual Health Questionnaire | 20 weeks
Davidson Sexual Encounter Profile | 20 weeks
Nocturnal penile tumescence and penile rigidity measures | 20 weeks
Prostate specific antigen | 20 weeks
Hematocrit | 20 weeks
Fasting lipid profile / atherogenic markers | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tapper J, Arver S, Pencina KM, Martling A, Blomqvist L, Buchli C, Li Z, Gagliano-Juca T, Travison TG, Huang G, Storer TW, Bhasin S, Basaria S. Muscles of the trunk and pelvis are responsive to testosterone administration: data from testosterone dose-response study in young healthy men. Andrology. 2018 Jan;6(1):64-73. doi: 10.1111/andr.12454. PMID 29280355
- [Derived] Bhasin S, Travison TG, Storer TW, Lakshman K, Kaushik M, Mazer NA, Ngyuen AH, Davda MN, Jara H, Aakil A, Anderson S, Knapp PE, Hanka S, Mohammed N, Daou P, Miciek R, Ulloor J, Zhang A, Brooks B, Orwoll K, Hede-Brierley L, Eder R, Elmi A, Bhasin G, Collins L, Singh R, Basaria S. Effect of testosterone supplementation with and without a dual 5alpha-reductase inhibitor on fat-free mass in men with suppressed testosterone production: a randomized controlled trial. JAMA. 2012 Mar 7;307(9):931-9. doi: 10.1001/jama.2012.227. PMID 22396515